CLINICAL TRIAL: NCT06330272
Title: Accuracy of Spectrophotometry in Determining the Mineralization of Molar-incisor Hypomineralization Lesions by CPP-ACPF Dental Mousse: Clinical Study
Brief Title: Accuracy of Spectrophotometry in Hypomineralized Lesions Treated With CPP-ACPF Dental Mousse: Clinical Study
Acronym: ASHLTDMCS
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Meire Coelho Ferreira (Other)
Collaborators: Fundação de Amparo à Pesquisa e Desenvolvimento Científico do Maranhão (Unknown)
Responsible Party: Sponsor-Investigator, Meire Coelho Ferreira, Principal Investigator, Universidade Ceuma
Organization: Universidade Ceuma (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UCeuma
Record Dates: First submitted 2024-03-19; First posted 2024-03-26 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Molar Incisor Hypomineralization
Keywords: molar hypomineralization; tooth mousse plus; tooth remineralization; data accuracy
MeSH Terms: conditions — Molar Hypomineralization

STUDY DESIGN:
Intervention Model Description: MIH lesions will receive prophylaxis with pumice stone before application of CPP-ACPF-based dental foam (Tooth Mousse PlusTM, GC Corporation, Tokyo, Japan).
  The application of Tooth Mousse Plus to the MIH lesion will be carried out under relative isolation and with the aid of a microbrush. The cream will remain on the surface for 1 minute. The application will be carried out once a week, for four consecutive weeks.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- CPP-ACPF treatment (Experimental): To apply the dental mousse, prophylaxis will first be carried out on teeth affected by pumice. The application of Tooth Mousse Plus to the MIH lesion will be carried out under relative isolation and with the aid of a microbrush, the amount of mousse will be a "pea grain". The cream will remain on the surface for 1 minute. The application will be carried out once a week, for four consecutive weeks.
  Interventions: Procedure: Application of dental mousse based on CPP-ACPF

INTERVENTIONS:
Procedure: Application of dental mousse based on CPP-ACPF — Treatment will begin with pumice prophylaxis of incisors with IMH lesions. After this step, the teeth will be dried before applying dental foam based on CPP-ACPF (Tooth Mousse PlusTM, GC Corporation, Tokyo, Japan).
  The application of Tooth Mousse PlusTM to the MIH lesion will be carried out under relative isolation and with the aid of a microbrush. The cream will remain on the surface for 1 minute, which will be timed. The application will be carried out once a week, for four consecutive weeks.

SUMMARY:
MIH is a condition with considerable prevalence in the child population. This structural defect, represented by a change in the color of the enamel, can be accompanied by structural loss and great sensitivity. Remineralizing agents have been used to strengthen compromised enamel. The objective of the study will be to measure the accuracy of a spectrophotometer (VITA Easyshade V) in determining the mineralization of IMH lesions by a CPP-ACPF dental mousse.

DETAILED DESCRIPTION:
Molar-incisor hypomineralization (MIH) is a qualitative structural defect of tooth enamel characterized by a marked opacity, asymmetrically involving the first permanent molars and incisors. Some products containing casein phosphopeptide-amorphous calcium phosphate fluoride (CPP-ACPF) have been used in children with MIH. Casein, a protein derived from milk, promotes a remineralizing effect through enzymes present in the oral cavity. The objective of the study will be to evaluate the accuracy of a spectrophotometer (VITA Easyshade V) in the indirect determination of the mineralization of IMH lesions by a dental foam based on CPP-ACPF (Tooth Mousse Plus™). Upper or lower permanent incisors of children aged 7 to 9 years will be included in the study. Two duly calibrated operators will select participants at the Ceuma University Pediatric Dentistry Clinic and the diagnosis of MIH lesions will be carried out using the European Association of Pediatric Dentistry (EAPD) criteria. Inclusion criteria will be permanent incisors with mild MIH lesions (marked opacities without structural loss) of at least 2mm in diameter, white or beige/yellowish in color and that do not present visible bacterial biofilm. Children with enamel malformation associated with syndromes, amelogenesis imperfecta, fluorosis and dental erosion will be excluded; and children allergic to milk proteins (casein). A questionnaire to collect demographic, socioeconomic information and etiological factors for MIH will be administered to parents/guardians. The color of the lesion will be measured before applying the dental foam at baseline and at other follow-up times. It will be measured using the VITA Easyshade V spectrophotometer (Vita Zahnfakrik, Bad Säckingen, Germany). This measurement will be represented by the luminosity parameter (L) and will occur three times on the same tooth to obtain the average values. The change in color (ΔL) of the lesion will be determined from the initial data minus the data after 1 month of evaluation (before the application of dental foam). The visual appearance of the lesion (opaque or shiny appearance) will be assessed initially (opaque lesion for inclusion of the tooth in the research) and further follow-up times (before applying the foam). The lesion will also be assessed tactilely (presence or absence of roughness) prior to the initial treatment and further follow-up times (before applying the foam). The presence of sensitivity will be assessed initially and during follow-up times (before applying the foam) using an air jet. Demographic, socioeconomic and data related to probable etiological factors for MIH will also be collected. The data will be subjected to descriptive and inferential analysis (tests for dependent measures and agreement analysis).

ELIGIBILITY:
Inclusion Criteria:

* Permanent incisors with mild MIH lesions (marked opacities without structural loss) of at least 2mm in diameter;
* White or beige/yellowish MIH lesions;
* Not present visible bacterial biofilm.

Exclusion Criteria:

* Children with enamel malformation associated with syndromes, amelogenesis imperfecta, fluorosis and dental erosion;
* Children allergic to milk proteins (casein).

Ages: 7 Years to 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 98 (Estimated)
Dates: Start 2025-05-15 (Actual); Primary Completion 2025-12-15 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
To measure the accuracy of a spectrophotometer (VITA Easyshade V) in determining the mineralization of IMH lesions by a CPP-ACPF dental mousse | 1 month
  The spectrophotometry analysis was determined by the Kappa statistic (95% confidence interval) (primary outcome of the study).

CONTACTS AND LOCATIONS:
Overall Officials: Meire C. Ferreira, PhD, Study Director — Uniceuma
Locations (1):
- Josue Montello, Universidade Ceuma, São Luís, Maranhão, Brazil

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Alaluusua S. Aetiology of Molar-Incisor Hypomineralisation: A systematic review. Eur Arch Paediatr Dent. 2010 Apr;11(2):53-8. doi: 10.1007/BF03262713. PMID 20403298
- [Background] Altan H, Yilmaz RE. Clinical evaluation of resin infiltration treatment masking effect on hypomineralised enamel surfaces. BMC Oral Health. 2023 Jul 3;23(1):444. doi: 10.1186/s12903-023-03140-6. PMID 37400849
- [Background] Americano GC, Jacobsen PE, Soviero VM, Haubek D. A systematic review on the association between molar incisor hypomineralization and dental caries. Int J Paediatr Dent. 2017 Jan;27(1):11-21. doi: 10.1111/ipd.12233. Epub 2016 Apr 21. PMID 27098755
- [Background] Aranha AC, Pimenta LA, Marchi GM. Clinical evaluation of desensitizing treatments for cervical dentin hypersensitivity. Braz Oral Res. 2009 Jul-Sep;23(3):333-9. doi: 10.1590/s1806-83242009000300018. PMID 19893971
- [Background] Bandeira Lopes L, Machado V, Botelho J, Haubek D. Molar-incisor hypomineralization: an umbrella review. Acta Odontol Scand. 2021 Jul;79(5):359-369. doi: 10.1080/00016357.2020.1863461. Epub 2021 Feb 1. PMID 33524270
- [Background] Baroni C, Marchionni S. MIH supplementation strategies: prospective clinical and laboratory trial. J Dent Res. 2011 Mar;90(3):371-6. doi: 10.1177/0022034510388036. Epub 2010 Dec 13. PMID 21149856
- [Background] Cardoso-Martins I, Pessanha S, Coelho A, Arantes-Oliveira S, Marques PF. Evaluation of the Efficacy of CPP-ACP Remineralizing Mousse in Molar-Incisor Hypomineralized Teeth Using Polarized Raman and Scanning Electron Microscopy-An In Vitro Study. Biomedicines. 2022 Dec 1;10(12):3086. doi: 10.3390/biomedicines10123086. PMID 36551842
- [Background] da Costa-Silva CM, Jeremias F, de Souza JF, Cordeiro Rde C, Santos-Pinto L, Zuanon AC. Molar incisor hypomineralization: prevalence, severity and clinical consequences in Brazilian children. Int J Paediatr Dent. 2010 Nov;20(6):426-34. doi: 10.1111/j.1365-263X.2010.01097.x. Epub 2010 Aug 24. PMID 20738434
- [Background] Dias CSCF, Giotto LM, Oliveira Favretto C. O Uso De Vernizes Fluoretados Nos Tratamentos De Hipersensibilidade Dentinária: Uma Abordagem Atual. Rev Saúde Multidiscip. 2022;11(1):20-5
- [Background] Fagrell TG, Dietz W, Jalevik B, Noren JG. Chemical, mechanical and morphological properties of hypomineralized enamel of permanent first molars. Acta Odontol Scand. 2010 Jul;68(4):215-22. doi: 10.3109/00016351003752395. PMID 20392131
- [Background] Bullio Fragelli CM, Jeremias F, Feltrin de Souza J, Paschoal MA, de Cassia Loiola Cordeiro R, Santos-Pinto L. Longitudinal Evaluation of the Structural Integrity of Teeth Affected by Molar Incisor Hypomineralisation. Caries Res. 2015;49(4):378-83. doi: 10.1159/000380858. Epub 2015 May 13. PMID 25998233
- [Background] Garot E, Rouas P, Somani C, Taylor GD, Wong F, Lygidakis NA. An update of the aetiological factors involved in molar incisor hypomineralisation (MIH): a systematic review and meta-analysis. Eur Arch Paediatr Dent. 2022 Feb;23(1):23-38. doi: 10.1007/s40368-021-00646-x. Epub 2021 Jun 24. PMID 34164793
- [Background] Jalevik B. Prevalence and Diagnosis of Molar-Incisor- Hypomineralisation (MIH): A systematic review. Eur Arch Paediatr Dent. 2010 Apr;11(2):59-64. doi: 10.1007/BF03262714. PMID 20403299
- [Background] Kumar A, Goyal A, Gauba K, Kapur A, Singh SK, Mehta SK. An evaluation of remineralised MIH using CPP-ACP and fluoride varnish: An in-situ and in-vitro study. Eur Arch Paediatr Dent. 2022 Feb;23(1):79-87. doi: 10.1007/s40368-021-00630-5. Epub 2021 May 31. PMID 34057698
- [Background] Olgen IC, Sonmez H, Bezgin T. Effects of different remineralization agents on MIH defects: a randomized clinical study. Clin Oral Investig. 2022 Mar;26(3):3227-3238. doi: 10.1007/s00784-021-04305-9. Epub 2021 Nov 25. PMID 34821978
- [Background] Rodd HD, Boissonade FM, Day PF. Pulpal status of hypomineralized permanent molars. Pediatr Dent. 2007 Nov-Dec;29(6):514-20. PMID 18254423
- [Background] Sezer B, Kargul B. Effect of Remineralization Agents on Molar-Incisor Hypomineralization-Affected Incisors: A Randomized Controlled Clinical Trial. J Clin Pediatr Dent. 2022 May 1;46(3):192-198. doi: 10.17796/1053-4625-46.3.4. PMID 35830636
- [Background] Soviero V, Haubek D, Trindade C, Da Matta T, Poulsen S. Prevalence and distribution of demarcated opacities and their sequelae in permanent 1st molars and incisors in 7 to 13-year-old Brazilian children. Acta Odontol Scand. 2009;67(3):170-5. doi: 10.1080/00016350902758607. PMID 19253064
- [Background] Weerheijm KL, Jalevik B, Alaluusua S. Molar-incisor hypomineralisation. Caries Res. 2001 Sep-Oct;35(5):390-1. doi: 10.1159/000047479. No abstract available. PMID 11641576
- [Background] Zawaideh FI, Owais AI, Mushtaha S. Effect of CPP-ACP or a Potassium Nitrate Sodium Fluoride Dentifrice on Enamel Erosion Prevention. J Clin Pediatr Dent. 2017;41(2):135-140. doi: 10.17796/1053-4628-41.2.135. PMID 28288296